CLINICAL TRIAL: NCT00200837
Title: Ethnopharmacological Studies in Oral Medicine
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: University of Illinois at Chicago (Other); Latin University of Costa Rica (Other)
Other Study IDs: K08AT000987-01 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-03-28 (Estimated); Status verified 2007-03

CONDITIONS: Oral Pain; Oral Ulcers; Oral Tumors
Keywords: oral mucosal pain; oral inflammations; anisillo; cordonsillo; Piperaceae; oral ulcers; oral tumors; mucosal pain; mucosal inflammations; cordoncillo
MeSH Terms: conditions — Oral Ulcer

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
These are ethnomedicine studies of plants used by rural and indigenous peoples for pain and oral inflammation relief.

DETAILED DESCRIPTION:
These are ethnomedicine studies of plants used by rural and indigenous peoples for pain relief in Central and South America.

ELIGIBILITY:
Inclusion Criteria:

* Patients who use plants to relieve oral pain, inflammations, ulcers, and tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-03; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Colvard, DDS, Principal Investigator — University of Illinois at Chicago
Locations (3):
- University of Illinois at Chicago, Chicago, Illinois, United States
- Universidad Nacional, Medellín, Colombia
- Universidad Latina de Costa Rica, San José, Costa Rica

REFERENCES:
- [Background] Colvard MD, Ashrafi SH, Alonge OK, Cordell GA. Smokeless tobacco-induced lamellar body abnormalities. Oral Dis. 2006 May;12(3):343-8. doi: 10.1111/j.1601-0825.2005.01211.x. PMID 16700746
- [Background] Alonge OK, Ashrafi SH, Colvard MD. Mitochondrial volume densities in the smokeless tobacco-treated hamster cheek pouch epithelium. Oral Dis. 2003 May;9(3):138-43. doi: 10.1034/j.1601-0825.2003.01814.x. PMID 12945595
- [Background] Colvard MD, Cordell GA, Villalobos R, Sancho G, Soejarto DD, Pestle W, Echeverri TL, Perkowitz KM, Michel J. Survey of medical ethnobotanicals for dental and oral medicine conditions and pathologies. J Ethnopharmacol. 2006 Aug 11;107(1):134-42. doi: 10.1016/j.jep.2006.04.005. Epub 2006 Apr 18. PMID 16735102
- [Background] Cordell GA, Colvard MD. Some thoughts on the future of ethnopharmacology. J Ethnopharmacol. 2005 Aug 22;100(1-2):5-14. doi: 10.1016/j.jep.2005.05.027. PMID 16009517
- See also: Mitochondrial volume densities in the smokeless tobacco-treated hamster cheek pouch epithelium. — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Abstract&list_uids=12945595&query_hl=1
- See also: Smokeless tobacco-induced lamellar body abnormalities. — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?CMD=search&DB=pubmed
- See also: Survey of medical ethnobotanicals for dental and oral medicine conditions and pathologies. — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?CMD=search&DB=pubmed
- See also: Some thoughts on the Future of Ethnopharmacology — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?CMD=search&DB=pubmed